CLINICAL TRIAL: NCT03277196
Title: A Phase 3, 2-Arm, Open-label Study to Evaluate the Safety and Pharmacodynamics of Long-term Ivacaftor Treatment in Subjects With Cystic Fibrosis Who Are Less Than 24 Months of Age at Treatment Initiation and Have an Approved Ivacaftor-Responsive Mutation
Brief Title: A Study to Evaluate the Safety of Long-term Ivacaftor Treatment in Participants With Cystic Fibrosis Who Are Less Than 24 Months of Age at Treatment Initiation and Have an Approved Ivacaftor-Responsive Mutation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VX15-770-126; 2017-001379-21 (EudraCT Number)
Record Dates: First submitted 2017-09-06; First posted 2017-09-08 (Actual); Results first posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ivacaftor Arm (Experimental): Participants less than (<) 24 months of age and weighing 5 to less than (<) 7 kilogram (kg) received 25 mg IVA every 12 hours (q12h), 7 to <14 kg received 50 mg IVA q12h, and those weighing 14 to <25 kg received 75 mg IVA q12h.
  Participants more than or equal (>=) 24 months of age and weighing <14 kg received 50 mg IVA q12h, and those weighing more than or equal to (>=)14 kg received 75 mg IVA q12h in the treatment period for up to 96 weeks.
  Doses were determined based on safety and pharmacokinetic (PK) data from parent study, age and weight.
  Interventions: Drug: IVA
- Observational Arm (No Intervention)

INTERVENTIONS:
Drug: IVA — Granules for oral administration.
  Other Names: VX-770; ivacaftor
  Arms: Ivacaftor Arm

SUMMARY:
This is a Phase 3, 2-arm, multicenter study with an open-label ivacaftor arm and an observational arm to evaluate the safety and efficacy of long-term ivacaftor treatment in participants with cystic fibrosis (CF) who are <24 months of age at treatment initiation and have an approved Ivacaftor-Responsive mutation.

ELIGIBILITY:
Inclusion Criteria:

Ivacaftor Arm: Participants From Study 124 (NCT02725567 ) Part B:

* Participants transitioning from Study 124 Part B must have completed the last study visit of Study 124 Part B.
* As judged by the investigator, parent or legal guardian must be able to understand protocol requirements, restrictions, and instructions; and must sign the informed consent form (ICF).

Ivacaftor Arm: Participants Not From Study 124 Part B:

* Confirmed diagnosis of CF, or 2 CF-causing mutations.
* An ivacaftor- responsive CFTR mutation on at least 1 allele. Participants will be eligible in countries/regions where ivacaftor is approved for use in participants 2 years of age and older.
* As judged by the investigator, parent or legal guardian must be able to understand protocol requirements, restrictions, and instructions; and must sign the ICF.

Observational Arm:

* Received ivacaftor treatment in Study 124 Part B and elected not to enroll or ineligible to enroll in the ivacaftor arm of Study 126.

Exclusion Criteria:

Ivacaftor Arm: Participants From Study 124 Part B:

* History of any illness or condition that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering ivacaftor to the participant.
* Participants receiving commercially available ivacaftor treatment

Ivacaftor Arm: Participants Not From Study 124 Part B:

* History of any illness or condition that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering ivacaftor to the participant
* An acute upper or lower respiratory infection, or pulmonary exacerbation, or changes in therapy for pulmonary disease within 4 weeks of Day 1
* Abnormal liver function at screening
* Hemoglobin <9.5 g/dL at screening
* History of solid organ or hematological transplantation
* Use of any moderate or strong inducers or inhibitors of CYP3A within 2 weeks of Day 1

Observational Arm:

* Receiving ivacaftor treatment

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 0 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-10-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - Alfred I DuPont Hospital for Children, Wilmington, Delaware
  - Nemours Children's Hospital, Orlando, Florida
  - Center for Advanced Pediatrics, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - John Hopkins Hospital, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Childrens's Hospitals and Clinics of Minnnesota, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Billings Clinic Hospital, Billings, Montana
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- Queensland Children's Hospital, South Brisbane, Australia
- The Hospital for Sick Children, Toronto, Ontario, Canada
- Universitaetsklinikum Heidelberg, Zenter fuer Kinder-und Jugendmedizin, Heidelberg, Germany
- Ireland (3):
  - Children's Health Ireland at Crumlin, Dublin
  - Children's University Hospital Temple Street, Dublin
  - University Hospital Limerick, Limerick
- United Kingdom (6):
  - Paediatric Clinical Research Facility, Edinburgh
  - Alder Hey Children's Alder Hey Children's NHS Foundation Trust, Liverpool
  - Great Ormond Street Hospital for Sick Children, London
  - Royal Brompton & Harefield NHS Founcation Trust, Royal BromptonHospital, London
  - Royal Manchester Children's Hospital, Manchester
  - Oxford University Hospitals NHS Trust, John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was planned to include 2 arms: an ivacaftor (IVA) arm (open-label, 96-week treatment period) and an observational arm. However, there were no participants enrolled in the observational arm. A total of 86 participants enrolled in the Ivacaftor arm.
Pre-assignment Details: Rollover participants (who completed parent study VX15-770-124 [NCT02725567] Part B or Part A/B) and IVA-naïve participants (who participated in study VX15-770-124 Part A only or who did not participate in VX15-770-124 and were less than (<) 24 months of age at the Day 1 of current study [VX15-770-126]) were enrolled in this study.
Groups:
- Ivacaftor Treatment: Participants less than (<) 24 months of age and weighing 5 to less than (<) 7 kilogram (kg) received 25 mg IVA every 12 hours (q12h), 7 to <14 kg received 50 mg IVA q12h, and those weighing 14 to <25 kg received 75 mg IVA q12h.
  Participants more than or equal (>=) 24 months of age and weighing <14 kg received 50 mg IVA q12h, and those weighing more than or equal to (>=)14 kg received 75 mg IVA q12h in the treatment period for up to 96 weeks.
Period: Overall Study
Arm/Group | Ivacaftor Treatment
Started | 86
Rollover Participants (Rollover Participants (who completed Study VX15-770-124 Part B or Part A/B).) | 38
IVA-Naïve Participants (IVA-naïve participants (who participated in study VX15-770-124 Part A only or who did not participate in VX15-770-124).) | 48 (A total of 86 participants were enrolled in the study. However, only 38 participants rolled over from the VX15-770-124 study Part B or Part A/B to this study, and the rest of the participants were enrolled in the IVA naive group. Participants in IVA naive group are those who participated in study VX15-770-124 Part A only or who did not participate in VX15-770-124.)
Completed | 58
Not Completed | 28
Not completed — Commercial Drug is Available for Participants | 20
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal of Consent (not due to AE) | 3
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Population: Baseline data was analyzed on safety Set which is defined as all participants who received at least 1 dose of study drug.
Groups:
- Ivacaftor Treatment: Participants <24 months of age and weighing 5 <7 kg received 25 mg IVA q12h, 7 to <14 kg received 50 mg IVA q12h, and those weighing 14 to <25 kg received 75 mg IVA q12h.
  Participants >=24 months of age and weighing <14 kg received 50 mg IVA q12h, and those weighing >=14 kg received 75 mg IVA q12h in the treatment period for up to 96 weeks.
Arm/Group | Ivacaftor Treatment
Number analyzed (Participants) | 86
Age, Continuous [Mean (Standard Deviation); unit: months] | 10.2 (5.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 79
  Not collected per local regulations | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 82
  Asian | 1
  Not collected per local regulations | 3

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability as Assessed by Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs
Time Frame: Day 1 up to Week 120
Population: Safety Set included all participants who received at least 1 dose of study drug in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Ivacaftor Treatment
Number analyzed (Participants) | 86
Participants
  Participants with TEAEs | 85
  Participants with SAEs | 21

2. Secondary Outcome: Absolute Change in Sweat Chloride
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Baseline at Week 96
Population: The Full Analysis Set (FAS) included all participants who were enrolled and have at least 1 post baseline efficacy assessment in this study. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome.
Measure: Mean (Standard Deviation); unit: millimole per liter (mmol/L)
Arm/Group | Ivacaftor Treatment
Number analyzed (Participants) | 33
millimole per liter (mmol/L) | -55.3 (25.0)

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 120
Description: Safety Set included all participants who received at least 1 dose of study drug in this study.
Groups:
- Ivacaftor Arm: Participants <24 months of age and weighing 5 <7 kg received 25 mg IVA q12h, 7 to <14 kg received 50 mg IVA q12h, and those weighing 14 to <25 kg received 75 mg IVA q12h.
  Participants >=24 months of age and weighing <14 kg received 50 mg IVA q12h, and those weighing >=14 kg received 75 mg IVA q12h in the treatment period for up to 96 weeks.
Arm/Group | Ivacaftor Arm
All-Cause Mortality (participants affected / at risk) | 0/86
Serious Adverse Events (participants affected / at risk) | 21/86
Other Adverse Events (participants affected / at risk) | 83/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ivacaftor Arm (N=86)
Adrenocortical insufficiency acute (Endocrine disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Bronchiolitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 9
Lower respiratory tract infection viral (Infections and infestations) | 1
Parainfluenzae virus infection (Infections and infestations) | 1
Periorbital cellulitis (Infections and infestations) | 1
Respiratory syncytial virus infection (Infections and infestations) | 1
Rhinovirus infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Viral rash (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Electrocardiogram QT shortened (Investigations) | 1
Electroencephalogram abnormal (Investigations) | 1
Pseudomonas test positive (Investigations) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Device dislocation (Product Issues) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ivacaftor Arm (N=86)
Constipation (Gastrointestinal disorders) | 13
Diarrhoea (Gastrointestinal disorders) | 15
Teething (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 22
Pyrexia (General disorders) | 34
Seasonal allergy (Immune system disorders) | 6
Conjunctivitis (Infections and infestations) | 9
Ear infection (Infections and infestations) | 19
Gastroenteritis (Infections and infestations) | 9
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 13
Influenza (Infections and infestations) | 8
Nasopharyngitis (Infections and infestations) | 10
Otitis media (Infections and infestations) | 10
Respiratory tract infection viral (Infections and infestations) | 5
Rhinitis (Infections and infestations) | 11
Sinusitis (Infections and infestations) | 6
Tonsillitis (Infections and infestations) | 6
Upper respiratory tract infection (Infections and infestations) | 24
Viral upper respiratory tract infection (Infections and infestations) | 6
Alanine aminotransferase increased (Investigations) | 7
Gamma-glutamyltransferase increased (Investigations) | 6
Haemophilus test positive (Investigations) | 6
Pseudomonas test positive (Investigations) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 60
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 13
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 33
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-10-05): https://cdn.clinicaltrials.gov/large-docs/96/NCT03277196/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-25): https://cdn.clinicaltrials.gov/large-docs/96/NCT03277196/SAP_001.pdf